CLINICAL TRIAL: NCT05528354
Title: Venetoclax and Decitabin Based Conditioning Regimen Followed With Post-HSCT Decitabin Maintenance Therapy in TP53 Mutant AML/MDS Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, He Huang, Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20220036C-R1
Record Dates: First submitted 2022-08-28; First posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Hematopoietic Stem Cell Transplantation; TP53
Keywords: hematopoietic stem cell transplantation; TP53; relapse; decitabine
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VEN and DEC based conditioning regimen followed with post-HSCT DEC maintenance therapy (Experimental)
  Interventions: Drug: VEN and DEC based conditioning regimen; Drug: DEC

INTERVENTIONS:
Drug: VEN and DEC based conditioning regimen — Patients with age<50 years and HCT-CI<3:
  Haploidentical transplantation: AraC 2g/m2 d-10~d-9, BU 0.8mg/kg q6h d-8~-6, CTX 1.8g/m2 d-5~d-4, Meccnu 250mg/m2 d-3, ATG 1.5mg/kg/d d-5~-2, VEN 400mg/d d-15~-9, DEC 20mg/m2 d-15~-11; HLA-matched transplantation: BU 0.8mg/kg q6h d-7~-4, CTX 60mg/kg d-3~d-2, Meccnu 250mg/m2 d-1, VEN d-12~-8, DEC 20mg/m2 d-12~-6, and ATG for the unrelated donor type.
  Patients with age>50 years or HCT-CI≥3:
  Flu 30mg/m2 d-10~-5, BU 0.8mg/kg q6h d-7~-5, Meccnu 250mg/m2 d-4, ATG 7.5mg/kg divided into d-4~-1, VEN d-15~-9, DEC 20mg/m2 d-15~-11.
  Note: if Voriconazole or Posaconazole is used to prevent or treat fungal infections, VEN should be 200mg/d for 7 consecutive days.
Drug: DEC — In the time window of 60-120 days after transplantation: DEC 5mg/m2/d for 5 consecutive days every 6 to 8 weeks with a total of 4 to 6 courses if there is no severe aGVHD (grade 3 or higher) and the donor chimerism rate of bone marrow blood (STR)>95%.
  If the MRD turns positive, DLI can be performed.

SUMMARY:
This study aims to evaluate the effectiveness and safety of Venetoclax and Decitabin based conditioning regimen followed with post-HSCT Decitabin maintenance therapy in TP53 mutant AML/MDS Patients.

DETAILED DESCRIPTION:
In acute myeloid leukemia and myelodysplastic syndromes, TP53 gene mutation is a poor prognostic factor and a strong indication for hematopoietic stem cell transplantation. However, because of the high relapse rate of myeloid tumors with TP53 mutation, new comprehensive treatment is urgently needed to improve the efficacy of transplantation. Decitabin(DEC) has shown certain efficacy in primary patients with TP53 mutation, and Venetoclax (VEN) and DEC have synergistic effect. Based on this, we hypothesized that DEC and VEN should be added to the conditioning regimen in TP53 mutant AML/MDS patients in order to eliminate malignant clones with P53 mutation as much as possible, and intermittent DEC maintenance therapy should be used to prevent relapse after post-HSCT hematopoietic reconstruction. We intend to conduct a multicenter, single-arm clinical study to evaluate the efficacy and safety of this protocol.

ELIGIBILITY:
Inclusion Criteria:

1. AML or MDS diagnosed according to 2016 WHO criteria with TP53 mutation before enrollment;
2. Aged from 12 to 70 years;
3. The Eastern Cooperative Oncology Group (ECOG) performance score of 0-2;
4. Creatinine clearance rate ≥ 60 mL/min (according to Cockcroft-Gault formula);
5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≥ 3× upper limit of normal range (ULN), total bilirubin ≤ 2×ULN;
6. Left ventricular ejection fraction (LVEF) assessed by echocardiography (ECHO) ≥ 45%;
7. Life expectancy > 8 weeks;
8. Sign the informed consent voluntarily, understand and comply with all trial requirements.

Exclusion Criteria:

1. Active autoimmune diseases, such as SLE, rheumatoid arthritis, etc.
2. Current active cardiovascular disease with clinically significance, such as uncontrolled arrhythmias, uncontrolled hypertension, congestive heart failure, any grade 3 or 4 heart disease determined by the New York Heart Association (NYHA) functional classification, or a history of myocardial infarction within the 6 months prior to screening;
3. Other serious medical conditions (e.g., advanced infection) that may limit the patient's participation in the trial;
4. Known human immunodeficiency virus (HIV) infection, or drug-uncontrolled chronic infection of hepatitis B virus (HBV-DNA > 1000IU/ml) or hepatitis C virus (anti-HCV positive);
5. Pregnant or lactating women;
6. Fail to understand, comply with the study protocol or sign the informed consent form.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | At Year 1
  The time from transplantation to the occurrence of any of the following:
  1. Death from any cause
  2. Disease recurrence, defined as one of the following:
  Leukemia blasts reappeared in peripheral blood, or blasts ≥ 5%, naive monocytes ≥ 5% in bone marrow, or extramedullary lesions.

SECONDARY OUTCOMES:
Overall survival (OS) | At Year 1
  Assessment of OS at Year 1
Cumulative relapse rate | At Year 1
  Assessment of cumulative relapse rate at Year 1
Non-relapse mortality (NRM) | At Year 1
  Assessment of NRM at Year 1
Acute graft-versus-host disease (GVHD) | At Day 100
  Acute GVHD incidence
Chronic graft-versus-host disease (GVHD) | through study completion, an average of 1 year
  Chronic GVHD incidence
Adverse effects | through study completion, an average of 1 year
  Drug related adverse effects

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Zhejiang Medical Colleage Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No